CLINICAL TRIAL: NCT01136655
Title: A Phase 2, Randomized, Blinded, 5-period Cross-over, Placebo and Active Controlled, Multicenter, Dose-finding Study Comparing Single Doses of Formoterol 2.25 µg, 4.5 µg, and 9 µg Delivered Via Symbicort pMDI and Foradil® 12 µg Evaluating the Relative Bronchodilating Effects and Safety in Children
Brief Title: A Study in Asthmatic Children (6 to <12 Yrs) Comparing Single Doses of Formoterol and Foradil® Evaluating Efficacy
Acronym: CHASE 2
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D589GC00002
Record Dates: First submitted 2010-06-01; First posted 2010-06-03 (Estimated); Results first posted 2013-08-30 (Estimated); Last update posted 2013-10-31 (Estimated); Status verified 2013-10

CONDITIONS: Asthma
Keywords: asthmatic children; Symbicort; Foradil
MeSH Terms: conditions — Asthma | interventions — Formoterol Fumarate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (5):
- BUD 160/FM 2.25 (Experimental): 2.25 μg formoterol (as 80/2.25 μg Symbicort pMDI × 1 inhalation) + 40 μg budesonide HFA pMDI × 2 inhalations
  Interventions: Drug: 80/2.25 μg Symbicort pMDI; Drug: 40 μg budesonide HFA pMDI
- BUD 160/FM 4.5 (Experimental): placebo HFA pMDI × 1 inhalation + 4.5 μg formoterol (as 80/2.25 μg Symbicort pMDI × 2 inhalations)
  Interventions: Drug: 80/2.25 μg Symbicort pMDI; Drug: placebo HFA pMDI
- BUD 160/FM 9.0 (Experimental): placebo HFA pMDI × 1 inhalation + 9 μg formoterol (as 80/4.5 μg Symbicort pMDI × 2 inhalations)
  Interventions: Drug: 80/4.5 μg Symbicort pMDI; Drug: placebo HFA pMDI
- BUD 160 (Placebo Comparator): placebo HFA pMDI × 1 inhalation + 80 μg budesonide HFA pMDI × 2 inhalations
  Interventions: Drug: 40 μg budesonide HFA pMDI; Drug: placebo HFA pMDI
- BUD 160/Foradil 12.0 (Active Comparator): Foradil Aerolizer 12 μg × 1 inhalation + 80 μg budesonide HFA pMDI × 2 inhalations
  Interventions: Drug: Foradil Aerolizer 12 μg; Drug: 40 μg budesonide HFA pMDI

INTERVENTIONS:
Drug: 80/2.25 μg Symbicort pMDI — inhalation
  Arms: BUD 160/FM 2.25; BUD 160/FM 4.5
Drug: 80/4.5 μg Symbicort pMDI — inhalation
  Arms: BUD 160/FM 9.0
Drug: Foradil Aerolizer 12 μg — inhalation
  Arms: BUD 160/Foradil 12.0
Drug: 40 μg budesonide HFA pMDI — inhalation
  Arms: BUD 160; BUD 160/FM 2.25; BUD 160/Foradil 12.0
Drug: placebo HFA pMDI — inhalation
  Arms: BUD 160; BUD 160/FM 4.5; BUD 160/FM 9.0

SUMMARY:
This purpose of the study is to investigate the bronchodilating effects of 3 different dosages of formoterol given in combination with budesonide as Symbicort pMDI.

DETAILED DESCRIPTION:
A Phase 2, randomized, blinded, 5-period cross-over, placebo and active controlled, multicenter, dose-finding study comparing single doses of formoterol 2.25 µg, 4.5 µg, and 9 µg delivered via Symbicort pMDI and Foradil® 12 µg evaluating the relative bronchodilating effects and safety in children.

ELIGIBILITY:
Inclusion Criteria:

* Has a documented clinical diagnosis of asthma for at least 6 months prior to Visit 1
* Has a FEV1 measured at least 6 hours after the last dose of inhaled, short-acting β2-agonist (SABA) and at least 48 hours after the last dose of inhaled long-acting β2-agonist of =60% and =85% of predicted normal.
* Demonstrated reversibility of FEV1 of =15% from pre short acting beta agonist level within 15 to 30 minutes after administration of a standard dose of short acting beta agonist

Exclusion Criteria:

* Has been hospitalized for >24 hours at least once or required emergency treatment or urgent care visit more than once for an asthma-related condition during the 6 months prior to Visit 1
* Has required treatment with systemic corticosteroids (eg, oral, parenteral, or rectal) for any reason within the 12 weeks prior to Visit 1.

Ages: 6 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 54 (Actual)
Dates: Start 2010-09; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lars-Goran Carlsson, MD, Study Director — AstraZeneca
Locations (34):
- United States (20):
  - Research Site, Huntington, California
  - Research Site, Long Beach, California
  - Research Site, Mission Viejo, California
  - Research Site, Orange, California
  - Research Site, Rolling Hills Estate, California
  - Research Site, Sarasota, Florida
  - Research Site, Omaha, Nebraska
  - Research Site, Morrisville, North Carolina
  - Research Site, Raleigh, North Carolina
  - Research Site, Eugene, Oregon
  - Research Site, Lake Oswego, Oregon
  - Research Site, Medford, Oregon
  - Research Site, Portland, Oregon
  - Research Site, Altoona, Pennsylvania
  - Research Site, Upland, Pennsylvania
  - Research Site, Charleston, South Carolina
  - Research Site, El Paso, Texas
  - Research Site, San Antonio, Texas
  - Research Site, Waco, Texas
  - Research Site, Springfield, Virginia
- Research Site, Dublin, Bulgaria
- Research Site, Dublin, Czechia
- Hungary (4):
  - Research Site, Budapest
  - Research Site, Dublin
  - Research Site, Miskolc
  - Research Site, Sopron
- Research Site, Dublin, Poland
- South Africa (7):
  - Research Site, Krugersdorp, Gauteng
  - Research Site, Pietermariztburg, KwaZulu-Natal
  - Research Site, Durban, Kz-natal
  - Research Site, Cape Town, South Africa
  - Research Site, Cape Town, W Cape
  - Research Site, Claremont, W Cape
  - Research Site, Dublin

REFERENCES:
- [Derived] Berger WE, Gillen M, Eckerwall G, Uryniak T, Trudo FJ, Lampl KL. Bronchodilator effect of single-dose formoterol administered by pressurized metered-dose inhaler in children with asthma aged 6 to <12 years receiving budesonide. Allergy Asthma Proc. 2014 Mar-Apr;35(2):134-40. doi: 10.2500/aap.2014.35.3746. PMID 24717790

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This multicenter study was conducted in Europe and the United States between 7 October 2010 and 3 January 2012.
Pre-assignment Details: The study consisted of a screening visit, an enrolment visit, a 1- to 2-week run-in (standardization) period, randomization at Visit 3, and 4 further visits (Visits 4-7)separated by approximately 7-day (minimum 3 days; maximum 14 days) wash-out (stabilization) periods. Subjects received 1 of 5 single-dose treatments at Visits 3-7, in random order.
Groups:
- Randomized Patients: All randomized patients
Period: BUD 160/FM 2.25 (1 Dose)
Arm/Group | Randomized Patients
Started | 54
Completed | 54
Not Completed | 0
Period: Washout After BUD 160/FM 2.25 (7 Days)
Arm/Group | Randomized Patients
Started | 54
Completed | 53
Not Completed | 1
Not completed — Withdrawal by Subject | 1
Period: BUD 160/FM 4.5 (1 Dose)
Arm/Group | Randomized Patients
Started | 53
Completed | 53
Not Completed | 0
Period: Washout After BUD 160/FM 4.5 (7 Days)
Arm/Group | Randomized Patients
Started | 53
Completed | 52
Not Completed | 1
Not completed — Adverse Event | 1
Period: BUD 160/FM 9.0 (1 Dose)
Arm/Group | Randomized Patients
Started | 53
Completed | 53
Not Completed | 0
Period: Washout After BUD 160/FM 9.0 (7 Days)
Arm/Group | Randomized Patients
Started | 53
Completed | 51
Not Completed | 2
Not completed — Withdrawal by Subject | 1
Not completed — Adverse Event | 1
Period: BUD 160 (1 Dose)
Arm/Group | Randomized Patients
Started | 51
Completed | 51
Not Completed | 0
Period: Washout After BUD 160 (7 Days)
Arm/Group | Randomized Patients
Started | 51
Completed | 51
Not Completed | 0
Period: BUD 160/ Foradil 12.0 (1 Dose)
Arm/Group | Randomized Patients
Started | 50
Completed | 50
Not Completed | 0
Period: Washout After BUD 160/ Foradil (7 Days)
Arm/Group | Randomized Patients
Started | 50
Completed | 50
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Randomized Patients
Number analyzed (Participants) | 54
Age Continuous [Mean (Standard Deviation); unit: years] | 9.2 (1.79)
Age, Customized [Number; unit: participants]
  >=6 to <8 years | 11
  >=8 to < 12 years | 43
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23
  Male | 31
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 22
  White | 31
  More than one race | 0
  Unknown or Not Reported | 1

OUTCOME MEASURES:

1. Primary Outcome: Average 12 Hour Forced Expiratory Volume in 1 Second (FEV1)
Description: Pulmonary function tests consisted of 3 forced expiratory maneuvers in which the patient expired forcefully from total lung capacity to residual volume, recorded using a spirometer. FEV1 was obtained from the full expiratory flow-volume-time curve. FEV1 was measured at 3, 9, 15, 60, 120, 180, 240, 360, 480, 600 and 720 minutes post administration of randomized study medication. Twelve-hour serial FEV1 was calculated through an AUC determination and then divided by time, so that the final value is expressed in liters. One subject was incorrectly administered BUD 160/ formoterol (FM) 9.0 rather than BUD 160/ Foradil 12.0 at Period 4. Hence this subject is included in the Efficacy Analysis Set, but not the Safety Analysis Set for BUD 160/ Foradil 12.0.
Time Frame: at 3, 9, 15, 60, 120, 180, 240, 360, 480, 600 and 720 minutes postdose
Population: Efficacy analysis set including all patients who were randomized (defined as having a randomization code recorded on the demography case report form), received at least one dose of study medication, and contributed sufficient data for at least one efficacy endpoint.
Measure: Least Squares Mean (Standard Error); unit: liters
Groups:
- BUD 160/FM 2.25: 2.25 μg formoterol (as 80/2.25 μg Symbicort pMDI x 1 inhalation) + 40 μg budesonide HFA pMDI × 2 inhalations
- BUD 160/FM 4.5: placebo HFA pMDI x 1 inhalation + 4.5 μg formoterol (as 80/2.25 μg Symbicort pMDI x 2 inhalations)
- BUD 160/FM 9.0: placebo HFA pMDI x 1 inhalation + 9 μg formoterol (as 80/4.5 μg Symbicort pMDI x 2 inhalations)
- BUD 160: placebo HFA pMDI x 1 inhalation + 80 μg budesonide HFA pMDI x 2 inhalations
- BUD 160/ Foradil 12.0: Foradil Aerolizer 12 μg x 1 inhalation + 80 μg budesonide HFA pMDI × 2 inhalations
Arm/Group | BUD 160/FM 2.25 | BUD 160/FM 4.5 | BUD 160/FM 9.0 | BUD 160 | BUD 160/ Foradil 12.0
Number analyzed (Participants) | 54 | 53 | 53 | 51 | 51
liters | 1.546 (0.0097) | 1.594 (0.0099) | 1.603 (0.0099) | 1.489 (0.0101) | 1.603 (0.0101)
Statistical Analysis 1: Comparison: BUD 160/FM 9.0 vs BUD 160; Factors in the ANCOVA model included: patient, visit, treatment, and the covariate pre-dose FEV1 from each visit; Test type: Superiority or Other; p < 0.0001, ANCOVA; LOCF was performed if missing data were post last non-missing post-baseline assessment; LS mean difference = 0.114, 95% CI 2-sided [0.087 to 0.142], Standard Error of Mean 0.0140
Statistical Analysis 2: Comparison: BUD 160/FM 4.5 vs BUD 160; Factors in the ANCOVA model included: patient, visit, treatment, and the covariate pre-dose FEV1 from each visit; Test type: Superiority or Other; p < 0.0001, ANCOVA; LOCF was performed if missing data were post last non-missing post-baseline assessment; LS mean difference = 0.105, 95% CI 2-sided [0.078 to 0.133], Standard Error of Mean 0.0140
Statistical Analysis 3: Comparison: BUD 160/FM 2.25 vs BUD 160; Factors in the ANCOVA model included: patient, visit, treatment, and the covariate pre-dose FEV1 from each visit; Test type: Superiority or Other; p = 0.0001, ANCOVA; LOCF was performed if missing data were post last non-missing post-baseline assessment; LS mean difference = 0.058, 95% CI 2-sided [0.030 to 0.085], Standard Error of Mean 0.0141
Statistical Analysis 4: Comparison: BUD 160/FM 4.5 vs BUD 160/FM 9.0; Factors in the ANCOVA model included: patient, visit, treatment, and the covariate pre-dose FEV1 from each visit; Test type: Superiority or Other; p = 0.5223, ANCOVA; LOCF was performed if missing data were post last non-missing post-baseline assessment; LS mean difference = -0.009, 95% CI 2-sided [-0.036 to 0.018], Standard Error of Mean 0.0139
Statistical Analysis 5: Comparison: BUD 160/FM 2.25 vs BUD 160/FM 9.0; Factors in the ANCOVA model included: patient, visit, treatment, and the covariate pre-dose FEV1 from each visit; Test type: Superiority or Other; p = 0.0001, ANCOVA; LOCF was performed if missing data were post last non-missing post-baseline assessment; LS mean difference = -0.057, 95% CI 2-sided [-0.084 to -0.029], Standard Error of Mean 0.0139
Statistical Analysis 6: Comparison: BUD 160/FM 2.25 vs BUD 160/FM 4.5; Factors in the ANCOVA model included: patient, visit, treatment, and the covariate pre-dose FEV1 from each visit; Test type: Superiority or Other; p = 0.0007, ANCOVA; LOCF was performed if missing data were post last non-missing post-baseline assessment; LS mean difference = -0.048, 95% CI 2-sided [-0.075 to -0.020], Standard Error of Mean 0.0138
Statistical Analysis 7: Comparison: BUD 160 vs BUD 160/ Foradil 12.0; Factors in the ANCOVA model included: patient, visit, treatment, and the covariate pre-dose FEV1 from each visit; Test type: Superiority or Other; p < 0.0001, ANCOVA; LOCF was performed if missing data were post last non-missing post-baseline assessment; LS mean difference = -0.114, 95% CI 2-sided [-0.142 to -0.086], Standard Error of Mean 0.0141
Statistical Analysis 8: Comparison: BUD 160/FM 2.25 vs BUD 160/ Foradil 12.0; Factors in the ANCOVA model included: patient, visit, treatment, and the covariate pre-dose FEV1 from each visit; Test type: Superiority or Other; p = 0.0001, ANCOVA; LOCF was performed if missing data were post last non-missing post-baseline assessment; LS mean difference = -0.056, 95% CI 2-sided [-0.084 to -0.028], Standard Error of Mean 0.0141
Statistical Analysis 9: Comparison: BUD 160/FM 4.5 vs BUD 160/ Foradil 12.0; Factors in the ANCOVA model included: patient, visit, treatment, and the covariate pre-dose FEV1 from each visit; Test type: Superiority or Other; p = 0.5394, ANCOVA; LOCF was performed if missing data were post last non-missing post-baseline assessment; LS mean difference = -0.009, 95% CI 2-sided [-0.036 to 0.019], Standard Error of Mean 0.0141
Statistical Analysis 10: Comparison: BUD 160/FM 9.0 vs BUD 160/ Foradil 12.0; Factors in the ANCOVA model included: patient, visit, treatment, and the covariate pre-dose FEV1 from each visit; Test type: Superiority or Other; p = 0.9863, ANCOVA; LOCF was performed if missing data were post last non-missing post-baseline assessment; LS mean difference = 0.000, 95% CI 2-sided [-0.027 to 0.028], Standard Error of Mean 0.0140

2. Secondary Outcome: FEV1 at 12 Hours After Study Medication Inhalation
Description: Pulmonary function tests consisted of 3 forced expiratory maneuvers in which the patient expired forcefully from total lung capacity to residual volume, recorded using a spirometer. The FEV1 value at 12 hours after dosing was taken as the 12-hour measurement (720 minutes) from the serial spirometry. One subject was incorrectly administered BUD 160/ formoterol (FM) 9.0 rather than BUD 160/ Foradil 12.0 at Period 4. Hence this subject is included in the Efficacy Analysis Set, but not the Safety Analysis Set for BUD 160/ Foradil 12.0.
Time Frame: 12 hours after dosing
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: liters
Arm/Group | BUD 160/FM 2.25 | BUD 160/FM 4.5 | BUD 160/FM 9.0 | BUD 160 | BUD 160/ Foradil 12.0
Number analyzed (Participants) | 54 | 53 | 53 | 51 | 51
liters | 1.641 (0.0175) | 1.692 (0.0177) | 1.731 (0.0177) | 1.626 (0.0181) | 1.709 (0.0182)
Statistical Analysis 1: Comparison: BUD 160/FM 9.0 vs BUD 160; Factors in the ANCOVA model included: patient, visit, treatment, and the covariate pre-dose FEV1 from each visit; Test type: Superiority or Other; p < 0.0001, ANCOVA; LOCF was performed if missing data were post last non-missing post-baseline assessment; LS mean difference = 0.105, 95% CI 2-sided [0.056 to 0.155], Standard Error of Mean 0.0250
Statistical Analysis 2: Comparison: BUD 160/FM 4.5 vs BUD 160; Factors in the ANCOVA model included: patient, visit, treatment, and the covariate pre-dose FEV1 from each visit; Test type: Superiority or Other; p = 0.0092, ANCOVA; LOCF was performed if missing data were post last non-missing post-baseline assessment; LS mean difference = 0.066, 95% CI 2-sided [0.017 to 0.116], Standard Error of Mean 0.0252
Statistical Analysis 3: Comparison: BUD 160/FM 2.25 vs BUD 160; Factors in the ANCOVA model included: patient, visit, treatment, and the covariate pre-dose FEV1 from each visit; Test type: Superiority or Other; p = 0.5509, ANCOVA; LOCF was performed if missing data were post last non-missing post-baseline assessment; LS mean difference = 0.015, 95% CI 2-sided [-0.035 to 0.065], Standard Error of Mean 0.0252
Statistical Analysis 4: Comparison: BUD 160/FM 4.5 vs BUD 160/FM 9.0; Factors in the ANCOVA model included: patient, visit, treatment, and the covariate pre-dose FEV1 from each visit; Test type: Superiority or Other; p = 0.1163, ANCOVA; LOCF was performed if missing data were post last non-missing post-baseline assessment; LS mean difference = -0.039, 95% CI 2-sided [-0.088 to 0.010], Standard Error of Mean 0.0249
Statistical Analysis 5: Comparison: BUD 160/FM 2.25 vs BUD 160/FM 9.0; Factors in the ANCOVA model included: patient, visit, treatment, and the covariate pre-dose FEV1 from each visit; Test type: Superiority or Other; p = 0.0004, ANCOVA; LOCF was performed if missing data were post last non-missing post-baseline assessment; LS mean difference = -0.090, 95% CI 2-sided [-0.140 to -0.041], Standard Error of Mean 0.0250
Statistical Analysis 6: Comparison: BUD 160/FM 2.25 vs BUD 160/FM 4.5; Factors in the ANCOVA model included: patient, visit, treatment, and the covariate pre-dose FEV1 from each visit; Test type: Superiority or Other; p = 0.0400, ANCOVA; LOCF was performed if missing data were post last non-missing post-baseline assessment; LS mean difference = -0.051, 95% CI 2-sided [-0.100 to -0.002], Standard Error of Mean 0.0247
Statistical Analysis 7: Comparison: BUD 160 vs BUD 160/ Foradil 12.0; Factors in the ANCOVA model included: patient, visit, treatment, and the covariate pre-dose FEV1 from each visit; Test type: Superiority or Other; p = 0.0011, ANCOVA; LOCF was performed if missing data were post last non-missing post-baseline assessment; LS mean difference = -0.083, 95% CI 2-sided [-0.133 to -0.034], Standard Error of Mean 0.0252
Statistical Analysis 8: Comparison: BUD 160/FM 2.25 vs BUD 160/ Foradil 12.0; Factors in the ANCOVA model included: patient, visit, treatment, and the covariate pre-dose FEV1 from each visit; Test type: Superiority or Other; p = 0.0077, ANCOVA; LOCF was performed if missing data were post last non-missing post-baseline assessment; LS mean difference = -0.068, 95% CI 2-sided [-0.118 to -0.018], Standard Error of Mean 0.0254
Statistical Analysis 9: Comparison: BUD 160/FM 4.5 vs BUD 160/ Foradil 12.0; Factors in the ANCOVA model included: patient, visit, treatment, and the covariate pre-dose FEV1 from each visit; Test type: Superiority or Other; p = 0.4957, ANCOVA; LOCF was performed if missing data were post last non-missing post-baseline assessment; LS mean difference = -0.017, 95% CI 2-sided [-0.067 to 0.033], Standard Error of Mean 0.0252
Statistical Analysis 10: Comparison: BUD 160/FM 9.0 vs BUD 160/ Foradil 12.0; Factors in the ANCOVA model included: patient, visit, treatment, and the covariate pre-dose FEV1 from each visit; Test type: Superiority or Other; p = 0.3800, ANCOVA; LOCF was performed if missing data were post last non-missing post-baseline assessment; LS mean difference = 0.022, 95% CI 2-sided [-0.027 to 0.071], Standard Error of Mean 0.0250

3. Secondary Outcome: Maximal FEV1 During the 12-hour Study Period
Description: Pulmonary function tests consisted of 3 forced expiratory maneuvers in which the patient expired forcefully from total lung capacity to residual volume, recorded using a spirometer. FEV1 was measured at 3, 9, 15, 60, 120, 180, 240, 360, 480, 600 and 720 minutes post administration of randomized study medication. The maximum FEV1 value was defined as the largest observed FEV1 value recorded during each 12-hour serial spirometry procedure. One subject was incorrectly administered BUD 160/ formoterol (FM) 9.0 rather than BUD 160/ Foradil 12.0 at Period 4. Hence this subject is included in the Efficacy Analysis Set, but not the Safety Analysis Set for BUD 160/ Foradil 12.0.
Time Frame: at 3, 9, 15, 60, 120, 180, 240, 360, 480, 600 and 720 minutes postdose
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: liters
Arm/Group | BUD 160/FM 2.25 | BUD 160/FM 4.5 | BUD 160/FM 9.0 | BUD 160 | BUD 160/ Foradil 12.0
Number analyzed (Participants) | 54 | 53 | 53 | 51 | 51
liters | 1.833 (0.0119) | 1.889 (0.0120) | 1.884 (0.0120) | 1.777 (0.0123) | 1.892 (0.0123)
Statistical Analysis 1: Comparison: BUD 160/FM 9.0 vs BUD 160; Factors in the Analysis of Covariance model included: patient, visit, treatment, and the covariate pre-dose FEV1 from each visit; Test type: Superiority or Other; p < 0.0001, ANCOVA; LS mean difference = 0.107, 95% CI 2-sided [0.073 to 0.140], Standard Error of Mean 0.0170
Statistical Analysis 2: Comparison: BUD 160/FM 4.5 vs BUD 160; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p < 0.0001, ANCOVA; LS mean difference = 0.112, 95% CI 2-sided [0.078 to 0.146], Standard Error of Mean 0.0171
Statistical Analysis 3: Comparison: BUD 160/FM 2.25 vs BUD 160; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.0011, ANCOVA; LS mean difference = 0.057, 95% CI 2-sided [0.023 to 0.090], Standard Error of Mean 0.0172
Statistical Analysis 4: Comparison: BUD 160/FM 4.5 vs BUD 160/FM 9.0; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.7589, ANCOVA; LS mean difference = 0.005, 95% CI 2-sided [-0.028 to 0.039], Standard Error of Mean 0.0169
Statistical Analysis 5: Comparison: BUD 160/FM 2.25 vs BUD 160/FM 9.0; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.0035, ANCOVA; LS mean difference = -0.050, 95% CI 2-sided [-0.084 to -0.017], Standard Error of Mean 0.0170
Statistical Analysis 6: Comparison: BUD 160/FM 2.25 vs BUD 160/FM 4.5; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.0011, ANCOVA; LS mean difference = -0.055, 95% CI 2-sided [-0.089 to -0.022], Standard Error of Mean 0.0168
Statistical Analysis 7: Comparison: BUD 160 vs BUD 160/ Foradil 12.0; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p < 0.0001, ANCOVA; LS mean difference = -0.115, 95% CI 2-sided [-0.149 to -0.081], Standard Error of Mean 0.0171
Statistical Analysis 8: Comparison: BUD 160/FM 2.25 vs BUD 160/ Foradil 12.0; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.0008, ANCOVA; LS mean difference = -0.058, 95% CI 2-sided [-0.092 to -0.024], Standard Error of Mean 0.0172
Statistical Analysis 9: Comparison: BUD 160/FM 4.5 vs BUD 160/ Foradil 12.0; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.8582, ANCOVA; LS mean difference = -0.003, 95% CI 2-sided [-0.037 to 0.031], Standard Error of Mean 0.0172
Statistical Analysis 10: Comparison: BUD 160/FM 9.0 vs BUD 160/ Foradil 12.0; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.6276, ANCOVA; LS mean difference = -0.008, 95% CI 2-sided [-0.042 to 0.025], Standard Error of Mean 0.0170

4. Secondary Outcome: Urinary Excretion of Formoterol During the 12 Hours Following Inhalation of Study Drug
Description: The amount of formoterol excreted unchanged in urine over the 12-hour period after administration [Ae(0-12h)] was calculated from the concentration of formoterol in urine multiplied by the total volume of urine collected. Volume was determined from the weight of the collected urine times an assumed urine density of 1020 g/L. The data for six patients who did not have measurable formoterol in their urine on the Foradil 12 μg treatment day was excluded from the analysis. All other urine concentrations below the lower limit of quantification were set to zero. One subject was incorrectly administered BUD 160/ formoterol (FM) 9.0 rather than BUD 160/ Foradil 12.0 at Period 4. Hence this subject is included in the Efficacy Analysis Set, but not the Safety Analysis Set for BUD 160/ Foradil 12.0.
Time Frame: 0 to 12 hours
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: pmol
Arm/Group | BUD 160/FM 2.25 | BUD 160/FM 4.5 | BUD 160/FM 9.0 | BUD 160/ Foradil 12.0
Number analyzed (Participants) | 51 | 52 | 51 | 43
pmol | 192.0 [156.36 to 235.88] | 366.3 [298.85 to 448.96] | 740.6 [602.45 to 910.51] | 658.7 [522.61 to 830.24]
Statistical Analysis 1: Comparison: BUD 160/FM 2.25 vs BUD 160/FM 4.5; Factors in the ANOVA model included: patient, period and treatment; Test type: Superiority or Other; p < 0.0001, ANOVA; A shift log transformation was performed on the response variable in the ANOVA model, using log(response) [log(response + 1) if response is 0]; LS mean difference = 0.52, 95% CI 2-sided [0.393 to 0.700]
Statistical Analysis 2: Comparison: BUD 160/FM 2.25 vs BUD 160/FM 9.0; Factors in the ANOVA model included: patient, period and treatment; Test type: Superiority or Other; p < 0.0001, ANOVA; [statistical method as in outcome 4, analysis 1]; LS mean difference = 0.26, 95% CI 2-sided [0.194 to 0.347]
Statistical Analysis 3: Comparison: BUD 160/FM 2.25 vs BUD 160/ Foradil 12.0; Factors in the ANOVA model included: patient, period and treatment; Test type: Superiority or Other; p < 0.0001, ANOVA; [statistical method as in outcome 4, analysis 1]; LS mean difference = 0.29, 95% CI 2-sided [0.214 to 0.396]
Statistical Analysis 4: Comparison: BUD 160/FM 4.5 vs BUD 160/FM 9.0; Factors in the ANOVA model included: patient, period and treatment; Test type: Superiority or Other; p < 0.0001, ANOVA; [statistical method as in outcome 4, analysis 1]; LS mean difference = 0.49, 95% CI 2-sided [0.371 to 0.659]
Statistical Analysis 5: Comparison: BUD 160/FM 4.5 vs BUD 160/ Foradil 12.0; Factors in the ANOVA model included: patient, period and treatment; Test type: Superiority or Other; p = 0.0002, ANOVA; [statistical method as in outcome 4, analysis 1]; LS mean difference = 0.56, 95% CI 2-sided [0.409 to 0.755]
Statistical Analysis 6: Comparison: BUD 160/FM 9.0 vs BUD 160/ Foradil 12.0; Factors in the ANOVA model included: patient, period and treatment; Test type: Superiority or Other; p = 0.4512, ANOVA; [statistical method as in outcome 4, analysis 1]; LS mean difference = 1.12, 95% CI 2-sided [0.827 to 1.528]

ADVERSE EVENTS:
Description: One subject was incorrectly administered BUD 160/ formoterol (FM) 9.0 rather than BUD 160/ Foradil 12.0 at Period 4. Hence this subject is included in the Efficacy Analysis Set, but not the Safety Analysis Set for BUD 160/ Foradil 12.0.
Arm/Group | BUD 160/FM 2.25 | BUD 160/FM 4.5 | BUD 160/FM 9.0 | BUD 160 | BUD 160/ Foradil 12.0
Serious Adverse Events (participants affected / at risk) | 0/54 | 0/53 | 0/53 | 0/51 | 0/50
Other Adverse Events (participants affected / at risk) | 1/54 | 1/53 | 5/53 | 2/51 | 0/50
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | BUD 160/FM 2.25 (N=54) | BUD 160/FM 4.5 (N=53) | BUD 160/FM 9.0 (N=53) | BUD 160 (N=51) | BUD 160/ Foradil 12.0 (N=50)
Headache (Nervous system disorders) | 1 | 1 | 5 | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days